CLINICAL TRIAL: NCT05166070
Title: An Exploratory Clinical Study to Evaluate the Safety and Efficacy of RD133 in Subjects With Relapsed or Refractory MSLN-Positive Solid Tumors
Brief Title: An Exploratory Clinical Study of RD133 in Subjects With Relapsed or Refractory MSLN-Positive Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Shanghai IASO Biotechnology Co., Ltd (Industry)
Responsible Party: Principal Investigator, Lingxiang Liu, Chief physician, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD133CI002
Record Dates: First submitted 2021-11-10; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Solid Tumor
Keywords: mesothelin-positive solid tumor; CAR-T

STUDY DESIGN:
Intervention Model Description: The study is a single center, open label, non-controlled, exploratory study. The "3+3"dose escalation design will be implemented to evaluate the safety and tolerability of RD133 in the treatment of subjects with relapsed/refractory MSLN-positive solid tumors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of RD133 (Experimental): Three dose groups of 1.0×10^6 CAR-T/kg, 3.0×10^6 CAR-T/kg, and 6.0×10^6 CAR-T/kg RD133 are designed in this study. 3 to 6 subjects are expected to be enrolled in each dose group according to observed DLT.
  RD133 will be intravenously infused at least 24 hours after lymphodepletion preconditioning. According to the assigned dose group, the designated dose of RD133 will be infused in a single infusion within 30 minutes on day 0.
  Interventions: Drug: RD133

INTERVENTIONS:
Drug: RD133 — The enhanced MSLN-CAR-T cell design of this study is obtained by co-infecting T cells with two lentiviral vectors. One lentiviral vector expresses CD19-CAR and tEGFR molecular safety switch, and the other lentiviral vector expresses MSLN- CAR and dnTGFβRII receptors. dnTGFβRII receptor without intracellular signal is used to resist the inhibition of T cell function by the immune microenvironment of tumor tissue. In addition, for the safety of CAR-T cell application in vivo, tEGFR is used in the CAR design as a molecular safety switch for CAR-T cells.

SUMMARY:
This study is a single-center exploratory clinical trial. It is estimated that 9-24 subjects will be enrolled. The "3+3" dose escalation design is adopted. The main purpose is to evaluate the safety of RD133 in the treatment of subjects with relapsed or refractory MSLN-positive solid tumors and explore the Recommend phase II dose of RD133 in the treatment of patients with relapsed/refractory MSLN-positive solid tumors.

DETAILED DESCRIPTION:
Leukapheresis procedure will be performed to manufacture RD133 chimeric antigen receptor (CAR) modified T cells. Bridging therapy is allowed between PBMC collection and lymphodepletion. Lymphodepletion with fludarabine and cyclophosphamide was performed for three consecutive days. After 1-day rest, subjects will receive a single dose infusion of RD133 at 1.0, 3.0, or 6.0x 10^6 CAR+ T cells/Kg. Subjects will be followed in the study for a minimum of 2 years after RD133 infusion. Long-term follow-up for lentiviral vector safety will be followed for up to 15 years after RD133 infusion.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must personally sign the written informed consent form approved by the ethics committee before the start of the study;
2. ≥18 years of age;
3. Have received at least 2 prior standard treatments, and achieved no response to the last-line treatment;
4. >25% Mesothelin positive rate on tumor cell membrane confirmed by prior immunohistochemistry of tumor tissue or freshly punctured tissue;
5. Expected survival ≥ 12 weeks;
6. ECOG score ≤ 2;
7. At least one measurable target lesion that meets the RECIST v1.1 standard;
8. Female or male subjects with fertility should agree to practice an effective method of contraception from the day of signing the ICF until 365 days after the infusion. Effective method of contraception is defined as: abstinence or contraceptive methods with an annual failure rate of <1% specified in the plan. ；
9. Before being enrolled in the group, the subject must have proper organ function and meet all of the following criteria:

9.1 The absolute value of neutrophils≥1.0×10^9/L (granulocyte colony stimulating factor (G-CSF) support is allowed, but must be without supportive treatment within 7 days before the examination); 9.2 Platelet count ≥75×10^9/L (must be without blood transfusion support [including blood component transfusion] or thrombopoietin [TPO], or other treatments for the purpose of increasing platelets within 7 days before the examination); 9.3 Hemoglobin ≥9 g/dl (must be without blood transfusion support [including blood component transfusion] within 7 days before the examination); 9.4 Bilirubin value ≤1.5×upper limit of normal (ULN) (except bile duct obstruction caused by tumor compression); 9.5 Creatinine clearance rate ≥60 ml/min; 9.6 ALT or AST ≤2.5×upper limit of normal (ULN) (with liver involvement ≤5×ULN); 9.7 The results of echocardiography indicate that the cardiac ejection fraction is ≥ 50%, without obvious pericardial effusion; 9.8 Stable coagulation function: INR ≤ 1.5, APTT ≤1.2×ULN (except tumor-related anticoagulation therapy); 9.9 >91% basic blood oxygen saturation in the natural indoor air environments.

Exclusion Criteria:

1. Subject who has received any of the following prior treatments:

   1.1 Subject with acute or chronic graft-versus-host disease (GVHD) who need systemic treatment within 4 weeks before enrollment; 1.2 Subject who has received gene therapy before enrollment; 1.3 Subject who needs systematic immunosuppressive therapy (except topical drugs) to control autoimmune diseases (eg: Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus, etc.), immunodeficiency or other diseases in the first 2 years after enrollment; 1.4 Subject who has been injected with live vaccines within 4 weeks before enrollment; 1.5 Subject has received other interventional clinical research drugs within 12 weeks before apheresis.
2. Subject with central metastasis or complete intestinal obstruction;
3. Subject with moderate or more severe hydrothorax and ascites which are hard to control by conventional treatment and require continuous catheter drainage;
4. With an active malignant tumor in the past 5 years, unless it is a curable tumor and has been obviously cured, such as basal or squamous cell carcinoma, cervical or breast carcinoma in situ, etc.
5. Subject with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and abnormal HBV DNA test results in peripheral blood (abnormal HBV DNA test results are defined as: HBV DNA quantitative level higher than the lower limit of the detection center or higher than normal range of the detection center; or qualitative HBV DNA test positive); Hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA positive; Human immunodeficiency virus (HIV) antibody positive; Cytomegalovirus ( CMV) DNA test positive; syphilis test RPR positive.
6. With an uncontrollable active infection (except genitourinary system infection and upper respiratory tract infection <CTCAE Grade 2).
7. Severe heart disease: including but not limited to unstable angina, myocardial infarction (within 6 months before screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ grade 3), severe arrhythmia.
8. Subject with hypertension that cannot be controlled by medication.
9. The toxicity of previous treatment has not been relieved to baseline or ≤1 (NCI-CTCAE v5.0, except for hair loss and laboratory abnormalities without clinical significance).
10. Major surgery within 2 weeks before enrollment, or has surgery planned during the time the subject is expected to be infused with RD133 or within 12 weeks after RD133 infusion (except planned surgery under local anesthesia).
11. Subject who has a solid organ transplant.
12. Women who are pregnant or breastfeeding.
13. Subject with previous central nervous system diseases (such as cerebral aneurysm, epilepsy, stroke, Alzheimer's disease, mental illness, etc.) or mental disorders.
14. Other unstable systemic diseases judged by the investigator: including but not limited to severe liver, kidney, or metabolic diseases that require medication.
15. Known to have life-threatening allergic reactions, hypersensitivity reactions or intolerances to RD133 cell preparations or its components.
16. Subject with hemorrhage, severe thrombosis judged by the Investigator, or hereditary/acquired hemorrhage and severe thrombosis (including hemophilia, coagulopathy, thrombocytopenia, hypersplenism, etc.), or are receiving thrombolytic or anticoagulant.
17. The researcher believes that other situations are not suitable for inclusion in the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2037-01-01 (Estimated)

PRIMARY OUTCOMES:
Type and incidence of dose-limiting toxicity (DLT) by dose group | 2 years post infusion
  The number and percentage of DLT in each dose group
Type and incidence of adverse events (AEs) and serious adverse events (SAEs) by dose group | 2 years post infusion
  Calculate type and incidence of adverse events (AE), serious adverse event (SAE), including those happened after lymphodepletion and after infusion, those related to study drug and lymphodepletion, or those that led to withdrawal from the study. They will also be aggregated by systematic organ classification (SOC), preferred term (PT), and severity.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events | 2 years post infusion
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product
Objective response rate (ORR) | 2 years post infusion
  The proportion of subjects who have achieved best response of partial response (PR) or complete response (CR) according to the RECIST V1.1 evaluation criteria 3 months after RD133 cell infusion.
Duration of response (DoR) | 2 years post infusion
  The time from the date of initial documentation of CR/PR after RD133 cell infusion to the date of progressive disease or death due to the disease studied
Time to response (TTR) | 2 years post infusion
  The time from the date of RD133 cell infusion to the first efficacy evaluation of partial response (PR) or complete response (CR)
Disease control rate (DCR) | 2 years post infusion
  The proportion of subjects with best efficacy assessment of complete response (CR), partial response (PR) or stable disease (SD)
Progression-free survival (PFS) | 2 years post infusion
  The time from the date of RD133 cell infusion to the date of initial documentation of progressive disease/relapse or death from any cause
Overall survival (OS) | 2 years post infusion
  The time from the date of RD133 cell infusion to the date of death
Transgene Levels of RD133 | 2 years post infusion
  Changes of virus vector copy number (VCN) in peripheral blood and tumor tissue (if any) after RD133 infusion
Chimeric Antigen Receptor T (CAR-T) Positive Cell Concentration | 2 years post infusion
  Changes of CAR T cell concentration in peripheral blood and tumor tissue (if any) after RD133 infusion

OTHER OUTCOMES:
Concentrations of TGF-β | 2 years post infusion
  Measurement of TGF-β level in peripheral blood
Expression of biomarker in tumor tissue | 2 years post infusion
  The expression of CD3, CD4, CD8, CD68, CD163, MSLN, and PDL1 in tumor tissue after RD133 cell infusion
Immunogenicity of RD133 | 2 years post infusion
  The positive rate and antibody level of human anti-RD133 antibodies after RD133 cell infusion
replication competent lentivirus (RCL) | 2 years post infusion
  The positive rate and change in replication competent lentivirus (RCL)
Exploratory analysis of MSLN level in peripheral blood | 2 years post infusion
  The correlation between MSLN level in peripheral blood before and after RD133 cell infusion
Exploratory analysis of MSLN level in tumor tissues and efficacy | 2 years post infusion
  The correlation between the expression level of MSLN in tumor tissues and clinical efficacy
T/B/NK cell ratio in peripheral blood | 2 years post infusion
  T/B/NK cell ratio in peripheral blood will be measured using flow cytometry after RD133 cell infusion
Systemic Cytokine Concentrations | 2 years post infusion
  Changes in the levels of inflammatory factors in peripheral blood after RD133 cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Lingxiang Liu, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No